CLINICAL TRIAL: NCT01320956
Title: Impact of Pre Operative Hypnosis on Anxiety in Children Aged 10 to 18 Years
Brief Title: Study of the Effects of Hypnosis Before Undergoing Surgery, on Anxiety in Children Aged 10 to 18 Years
Acronym: HYPOPANX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: P100112; 2010-A01165-34 (Other: ID-RCB)
Record Dates: First submitted 2011-03-21; First posted 2011-03-23 (Estimated); Last update posted 2023-02-06 (Actual); Status verified 2013-09

CONDITIONS: Osteotomy and Spinal Column Surgery
Keywords: hypnosis; HYPNOANALGESIA; surgery; children; anxiety; morphine; pain; A-VAS; orthopaedics; osteotomy; tenotomy; arthrodesis; spinal column surgery
MeSH Terms: conditions — Anxiety Disorders; Pain; Ankylosis | interventions — Hypnosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypnosis (Experimental): Pre operative nurse consultation and Hypnosis:
  will have hypnosis
  Interventions: Behavioral: Pre operative nurse consultation and Hypnosis
- Control (Active Comparator): Pre operative nurse consultation:
  usual nurse consultation without hypnosis
  Interventions: Other: Pre operative nurse consultation

INTERVENTIONS:
Behavioral: Pre operative nurse consultation and Hypnosis — Pre operative nurse consultation with pain management nurse, the day before surgery and 5 to 10 minutes of hypnosis, just before anesthesia, with trained nurse.
  Other Names: Hypnosis, HYPNOANALGESIA
  Arms: Hypnosis
Other: Pre operative nurse consultation — Pre operative nurse consultation with pain management nurse. Usual care and anesthesia
  Other Names: Control
  Arms: Control

SUMMARY:
This study aims to find how hypnosis performed just before a painful surgery can change anxiety level, in children aged 10 to 18 years.

DETAILED DESCRIPTION:
Undergoing surgery can cause anxiety among children. Thus, peri operative anxiety can increase levels of pain, need for painkillers, and even length of stay in hospital.

Caring for children must take in account their anxiety. This anxiety can be treated through drugs or others means such as hypnosis. Thus, the use hypnosis in surgery has been very poorly assessed.

Parents will be given a consent form as well as an information note. This study aims to compare the level of post operative anxiety (D1)of children having hypnosis before receiving anaesthetics to the level of anxiety of children getting the usual care.

All the children included in this study will have a pre operative consultation with the Pain Management Nurse.

The study applies to inpatients, aged 10 to 18 years, who must go through orthopaedics surgery such as osteotomy (bone section) and spinal column surgery. 120 patients will be included in this study (60 in each arm) The primary outcome measure is the level of anxiety at day 1 (24 hours after surgery) Other outcome measure are

* the difference in anxiety level between D-1 (the day before surgery) and D1 (24 hours after surgery)
* the use of morphine during the first 24 hours This study is a prospective randomized trial, comparing a usual analgesics procedure to an experimental analgesics procedure including hypnosis before anaesthesia.

Expected impact of this study :change in procedures, decrease of anxiety levels in patients by the use of hypnosis before anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* age 10-18 years
* Orthopaedics surgery (spinal column, osteotomy)
* ASA 1 & 2

Exclusion Criteria:

* casualty surgery
* patient or family unable to understand the study (language, disability ...)
* patient or family refusing the study

Ages: 10 Years to 215 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2011-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Level of anxiety at day 1 (24 hours after surgery) | 24 hours
  Level anxiety will be measured 24 hours after exit of operating room, using A-VAS (Anxiety visual analog scale) by a single blind assessor.

SECONDARY OUTCOMES:
Anxiety level | 24 hours
  difference in anxiety level between D-1 (the day before surgery) and D1 (24 hours after surgery)
Pain after surgery | 24 hours
  need for analgesics (morphine)

CONTACTS AND LOCATIONS:
Overall Officials: Chantal WOOD, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Robert Debré, Paris, France

REFERENCES:
- [Result] Duparc-Alegria N, Tiberghien K, Abdoul H, Dahmani S, Alberti C, Thiollier AF. Assessment of a short hypnosis in a paediatric operating room in reducing postoperative pain and anxiety: A randomised study. J Clin Nurs. 2018 Jan;27(1-2):86-91. doi: 10.1111/jocn.13848. Epub 2017 Jul 4. PMID 28403569